CLINICAL TRIAL: NCT04308694
Title: A Pilot Study to Permit Opioid Treatment Program Physicians to Prescribe Methadone Through Community Pharmacies for Their Stable Methadone Patients
Brief Title: Opioid Treatment Program (OTP)-Pharmacy Collaboration for Methadone Maintenance Treatment
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: Duke Health (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00103270; 3U01DA046910-02S3 (NIH)
Record Dates: First submitted 2020-03-10; First posted 2020-03-16 (Actual); Results first posted 2021-12-02 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pharmacy-based methadone treatment (Experimental): Participants will have their usual methadone dose administered and dispensed at a participating pharmacy. All other methadone services including counseling, drug testing, and medical services will be delivered as usual at the Methadone Program.
  Interventions: Drug: Pharmacy-based methadone administration and dispensing

INTERVENTIONS:
Drug: Pharmacy-based methadone administration and dispensing — Eligible participants receiving between 6- and 13-days of methadone take-home doses will have methadone administration and dispensing transferred from the opioid treatment program to the partnered community pharmacy. Each participant will be assessed monthly for 3 months (at 1, 2, and 3 months following intake/baseline) to explore the feasibility of transferring their methadone administration and dispensing to the select community pharmacy.

SUMMARY:
The overarching goal of this pilot study is to explore the feasibility, acceptability, and patient/provider satisfaction of pharmacy-based administration and dispensing of methadone for opioid use disorder. The results gained will inform the development of a future multisite randomized clinical trial.

DETAILED DESCRIPTION:
The study will use a non-randomized, prospective, single group design. Twenty long-term, clinically-stable methadone maintenance treatment (MMT) patients who receive between 6- and 13-days methadone take-home doses will be enrolled in the study where their methadone take-home administration and dispensing will be transferred to a community pharmacy for 3 months. Participants will also complete three follow-up assessments at 1-month, 2-months, and 3-months after the baseline visit to collect clinical and safety information since the previous assessment. Primary outcomes will be focused on feasibility measures (recruitment, accessibility to methadone treatment, substance use, medication call back success, and retention in treatment). Secondary outcomes will be focused on self-reported satisfaction measures from MMT providers (e.g., physician, physician assistant, nurse, and counselor) pharmacists, and patient participants.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or older receiving methadone treatment at Morse Clinic in Raleigh or Zebulon, NC.
* Able to provide informed written consent to participate in the pilot study.
* Receiving a stable methadone dose between 5 mg and 160 mg.
* Having all negative drug tests (except for prescribed methadone and ethanol) at the OTP for the past 12 months.
* No missed call-backs in the past 12 months.
* No signs/symptoms of a co-occurring major mental illness (i.e., thought disorder, thoughts of harm to self or others, delusions or hallucinations, cognitive impairment compromising informed consent to study procedures and requirements).
* Meeting the federal and state regulations for eligibility to receive between 6- and 13-days of take-home methadone and receiving this level of take-home doses at the time of study enrollment.
* If female, using adequate birth control methods.

Exclusion Criteria:

* Have a serious medical, psychiatric or substance use disorder that, in the opinion of the study physician, would make study participation hazardous to the participant, compromise study findings, or prevent the participant from completing the study.
* Have chronic pain requiring ongoing pain management with opioid analgesics.
* Prisoner status or pending legal action that could prevent participation in study activities
* Legal order for treatment (e.g., parole, probation, or pre-trial)
* Pregnant or breastfeeding at the time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzy Wu, ScD, Principal Investigator — Duke Health
Locations (3):
- United States (3):
  - Health Park Pharmacy, Raleigh, North Carolina
  - Morse Clinic of North Raleigh, Raleigh, North Carolina
  - Morse Clinic of Zebulon, Zebulon, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu LT, John WS, Morse ED, Adkins S, Pippin J, Brooner RK, Schwartz RP. Opioid treatment program and community pharmacy collaboration for methadone maintenance treatment: results from a feasibility clinical trial. Addiction. 2022 Feb;117(2):444-456. doi: 10.1111/add.15641. Epub 2021 Aug 16. PMID 34286886

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pharmacy-based Methadone Treatment
Started | 20
Completed | 16
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Pharmacy-based Methadone Treatment
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Rate
Description: The recruitment rate will be assessed on a monthly basis (e.g, Month 1, 2 and 3) until the enrollment target is reached. The recruitment rate is operationalized as the total number of participants consented in one month.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacy-based Methadone Treatment
Number analyzed (Participants) | 20
Participants
  Month 1 | 3
  Month 2 | 12
  Month 3 | 5

2. Primary Outcome: Treatment Adherence
Description: Adherence to pharmacy-based methadone treatment will be defined as the percentage of methadone take-home doses dispensed at the pharmacy out of the total number of take home doses prescribed.
Time Frame: Up to 3 months per participant
Population: All participants who began pharmacy-based methadone treatment.
Measure: Number; unit: percentage of dose adherence
Arm/Group | Pharmacy-based Methadone Treatment
Number analyzed (Participants) | 20
percentage of dose adherence | 100

3. Primary Outcome: Treatment Retention
Description: Treatment retention will be determined by the percentage of participants who remain in treatment at the pharmacy during the 3-month follow-up phase.
Time Frame: Up to 3 months per participant
Measure: Number; unit: percentage of participants retained
Arm/Group | Pharmacy-based Methadone Treatment
Number analyzed (Participants) | 20
percentage of participants retained | 80

4. Primary Outcome: Opioid and Other Substance Use
Description: The percentage of positive urine drug screens over the study duration will be examined.
Time Frame: Up to 3 months per participant
Population: A total of 52 urine drug tests were analyzed for the 20 participants enrolled in the study.
Measure: Number; unit: Percentage of positive tests
Units Other Than Participants: Urine Drug Tests
Arm/Group | Pharmacy-based Methadone Treatment
Number analyzed (Participants) | 20
Number analyzed (Urine Drug Tests) | 52
Percentage of positive tests | 3.8

5. Secondary Outcome: Treatment Satisfaction
Description: Participant satisfaction with treatment delivery will be measured on a monthly basis and a percentage of overall monthly ratings (combined) of satisfied or very satisfied will be calculated.
Time Frame: Over 3 months of treatment
Measure: Number; unit: percentage of satisfied ratings
Arm/Group | Pharmacy-based Methadone Treatment
Number analyzed (Participants) | 16
percentage of satisfied ratings | 87.5

6. Secondary Outcome: Adverse Events
Description: We will measure the prevalence of any fatal or non-fatal substance-related overdose and any substance-related emergency department visit or hospitalization.
Time Frame: Up to 3 months per participant
Measure: Number; unit: percentage
Arm/Group | Pharmacy-based Methadone Treatment
Number analyzed (Participants) | 20
percentage
  % of fatal and non-fatal overdoses | 0
  % of substance-related emergency department visits or hospitalizations | 0

7. Secondary Outcome: Percentage of Participants With Methadone Call Backs With Evidence of Tampering.
Description: Percentage of participants with call backs with evidence of methadone tampering.
Time Frame: 3 months
Population: Participants who had methadone call back.
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacy-based Methadone Treatment
Number analyzed (Participants) | 17
Participants | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Pharmacy-based Methadone Treatment
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pharmacy-based Methadone Treatment (N=20)
Non-study related hospitalization for abdominal pain (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/94/NCT04308694/Prot_SAP_000.pdf